CLINICAL TRIAL: NCT00935467
Title: A Study to Characterize the Steady-State Pharmacokinetics and Pharmacodynamics of 2.5 mg Saxagliptin Administered Twice Daily With Meals to Healthy Subjects
Brief Title: Pharmacokinetics and Pharmacodynamics Study of Saxagliptin in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CV181-091
Record Dates: First submitted 2009-07-08; First posted 2009-07-09 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-05

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — saxagliptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Saxagliptin (Other)
  Interventions: Drug: Saxagliptin

INTERVENTIONS:
Drug: Saxagliptin — Tablets, oral, 2.5 mg, twice daily, 7 days
  Other Names: Onglyza™

SUMMARY:
To characterize the steady-state pharmacokinetics (PK) of 2.5 mg saxagliptin administered twice daily with meals to healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* Men and women ages 18 to 45 inclusive
* Healthy subjects as determined by no clinically significant deviation from normal in medical history, physical examination, ECGs, and clinical laboratory determinations
* Body Mass Index (BMI) of 18 to 32 kg/m², inclusive. BMI = weight (kg)/ [height (m)]²

Exclusion Criteria:

* WOCBP who are unwilling or unable to use acceptable barrier methods (condoms and spermicides) to avoid pregnancy for the entire study period and for up to 8 weeks after the last dose of investigational product
* Any significant acute or chronic medical illness
* Current or recent (within 3 months) gastrointestinal disease
* Any major surgery within 4 weeks of study drug administration
* History of allergy to DPP4 inhibitor or related compounds
* Prior exposure to saxagliptin

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2009-07; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Evidence of steady-state pharmacokinetics (PK) of 2.5 mg saxagliptin administered twice daily with meals to healthy subjects | Within the first 24 hours of dosing

SECONDARY OUTCOMES:
To characterize the steady-state pharmacodynamics of 2.5 mg saxagliptin administered twice daily with meals to healthy subjects | 18 time points up to 14 hours on two separate study days
To assess the PK of the pharmacologically active major metabolite of saxagliptin, BMS-510849, following administration of 2.5 mg saxagliptin twice daily with meals to healthy subjects | 21 time points up to 23 hours after first dosing
To assess the safety and tolerability of 2.5 mg saxagliptin administered twice daily with meals to healthy subjects | Day 1 to Day 7

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Ppd Development, Lp, Austin, Texas, United States

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx